CLINICAL TRIAL: NCT00382707
Title: Transcranial Magnetic Stimulation and Anti-epileptic Effect: Optimization and Evaluation With Electrophysiology.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Premature termination following the departure of the principal investigator. No replacement investigator. Management decision.
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3540
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Refractory Frontal Lobe Epilepsy
Keywords: repetitive transcranial magnetic stimulation; low frequency; frontal lobe epilepsy; brain excitability; electromyography
MeSH Terms: conditions — Epilepsy, Frontal Lobe

INTERVENTIONS:
Device: cortical magnetic stimulation provided by an eight-shaped coïl placed upon the skull.

SUMMARY:
Epileptic disease is characterised by enhanced brain excitability. Low frequency repetitive transcranial magnetic stimulation (rTMS) can be an effective treatment for refractory frontal epilepsy. Thought, physiological mechanisms of its effectivity are still unknown. It is yet possible to evaluate cortical excitability and inhibition with TMS-coupled electromyography before and after rTMS sessions ; this could provide clues for basic mechanisms of rTMS effects on the epileptic brain. We assume that rTMS decrease brain excitability by improving brain inhibition. Such an information could help for treating patients with both pharmacological and non-pharmacological methods.

ELIGIBILITY:
Inclusion Criteria:

* Cryptogenic frontal lobe epilepsy
* Normal cerebral MRI

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2006-05 (Actual); Primary Completion 2009-09-01 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Electrophysiological parameters for cortical excitability measured just before and after rTMS, 4 hours later and 24 hours later.

SECONDARY OUTCOMES:
Clinical efficacity on seizure intensity and frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Serge CHASSAGNON, MD, Study Director — Hôpitaux Universitaires de Strasbourg
Locations (2):
- France (2):
  - Département de Neurologie - Hôpital Civil, Strasbourg
  - Institut de Physique Biologique, Strasbourg